CLINICAL TRIAL: NCT02665299
Title: Determination of the Utility of Plasma Circulating Tumor DNA (ctDNA) Measurements for the Detection of Colon Cancer in Patients Undergoing Diagnostic Colonoscopy
Brief Title: Plasma ctDNA in Patients Undergoing Diagnostic Colonoscopy
Status: Completed | Type: Observational
Sponsor: Pathway Genomics (Industry)
Responsible Party: Sponsor
Other Study IDs: Pathway Genomics 005
Record Dates: First submitted 2016-01-22; First posted 2016-01-27 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Colon Cancer; Colon Adenomas; Colon Polyps
Keywords: colon cancer; colon polyps; colon adenomas; colonoscopy; circulating tumor DNA
MeSH Terms: conditions — Colonic Neoplasms; Colonic Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood is drawn and DNA is purified from the plasma. The DNA is analyzed for circulating tumor DNA. The DNA will be stored for up to 10 years.
Oversight: Data Monitoring Committee: No

SUMMARY:
When the DNA inside of human cells undergoes certain alterations (mutations), the cells may develop into a cancer. The cancer cells may shed this DNA into the blood stream. This circulating tumor DNA (ctDNA) can be detected by very sensitive, specialized laboratory tests. Measurement of ctDNA has been shown to be useful for following patients with known cancer. It has also been found in the circulation of some patients with early stage cancer. The purpose of this study is to examine blood specimens for the presence of ctDNA in individuals without known cancer who are scheduled to undergo a screening or diagnostic colonoscopy in order to see if the ctDNA test can detect a cancer or precancerous condition at a very early stage before the patient becomes symptomatic. The results of this study should help define the role of ctDNA in the detection of early stage colon cancer and to define how sensitive it is (i.e. how well it picks up cancer when it is present) and how specific it is (i.e. how often is ctDNA found in patients with benign diseases or no abnormalities).

DETAILED DESCRIPTION:
After the participants have undergone the informed consent process, they will have 30 milliliters (approximately two tablespoons) of blood drawn. This will be done prior to their scheduled screening or diagnostic colonoscopy. If the patient has indicated a desire to receive the results of their test, they will receive a written description, as will their primary care physician. The patients will be contacted yearly for up to 5 years by the study staff to learn whether they have been found to have a diagnosis of colon or other cancer.

ELIGIBILITY:
Inclusion Criteria: .

* 18 years of age or older who are scheduled to undergo a screening or diagnostic colonoscopy by Dr. Phillip Fleshner

Exclusion Criteria:

* Prior history of cancer excluding basal cell carcinoma of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals 18 years of age or older without a prior diagnosis of cancer who are scheduled to undergo a screening or diagnostic colonoscopy by Dr. Phillip Fleshner.
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2016-01; Primary Completion 2017-04 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Utility of plasma ctDNA measurements to detect colon cancer or precancerous conditions. | 1 year
  Correlation between plasma ctDNA results and any pathology found at time of diagnostic colonoscopy. Determination of true positive, false positive and predictive values for using ctDNA measurements to detect colon cancer and precancerous conditions.

SECONDARY OUTCOMES:
Determination of incident rate of new colon or other cancers in patients who underwent initial measurement of ctDNA | 5 years
  Subjects will be contacted yearly to obtain follow-up information regarding the development of colon or other cancer in order to see if the initial ctDNA measurement detected the cancer before it became clinically apparent.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn D Braunstein, MD, Principal Investigator — Pathway Genomics
Locations (1):
- Pathway Genomics, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with the participants and their primary care physician

REFERENCES:
- [Background] Perrone F, Lampis A, Bertan C, Verderio P, Ciniselli CM, Pizzamiglio S, Frattini M, Nucifora M, Molinari F, Gallino G, Gariboldi M, Meroni E, Leo E, Pierotti MA, Pilotti S. Circulating free DNA in a screening program for early colorectal cancer detection. Tumori. 2014 Mar-Apr;100(2):115-21. doi: 10.1177/030089161410000201. PMID 24852853